CLINICAL TRIAL: NCT03792555
Title: A Double-blind, Placebo-controlled, Randomized Withdrawal Study to Evaluate the Safety, Pharmacokinetics and Efficacy of CRN00808 in Patients With Acromegaly That Are Responders to Octreotide LAR or Lanreotide Depot (ACROBAT Evolve)
Brief Title: A Study to Evaluate the Safety and Efficacy of Paltusotine for the Treatment of Acromegaly (ACROBAT Evolve)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Crinetics Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CRN00808-02; 2018-001833-42 (EudraCT Number)
Record Dates: First submitted 2018-12-27; First posted 2019-01-03 (Actual); Results first posted 2025-03-17 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Acromegaly
Keywords: Acromegaly; ACROBAT; EVOLVE; Paltusotine
MeSH Terms: conditions — Acromegaly

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Paltusotine (Experimental)
  Interventions: Drug: Paltusotine
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Paltusotine — Paltusotine, capsules, once daily by mouth
  Other Names: CRN00808
  Arms: Paltusotine
Drug: Placebo — Placebo, capsules, once daily by mouth
  Arms: Placebo

SUMMARY:
A Phase 2 double-blind, placebo-controlled, randomized withdrawal study is designed to evaluate the safety, efficacy, and pharmacokinetics of paltusotine (formerly CRN00808) in subjects with acromegaly that are responders to octreotide LAR or lanreotide depot.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects 18 to 75 years of age
2. Confirmed diagnosis of acromegaly that is controlled on stable doses of octreotide LAR or lanreotide depot
3. Females must be non-pregnant and non-lactating, and either surgically sterile, post-menopausal, or using effective method(s) of birth control
4. Willing to provide signed informed consent

Exclusion Criteria:

1. Treatment naïve acromegaly subjects
2. Prior treatment with paltusotine
3. Pituitary surgery within 6 months prior to Screening or radiation therapy at any time prior to the study entry. Pituitary radiation therapy (within 3 to 4 years or more than 4 years prior to study entry) with recently documented elevated IGF-1 may be eligible.
4. History or presence of malignancy except adequately treated basal cell and squamous cell carcinomas of the skin within the past 5 years.
5. Use of any investigational drug within the past 30 days or 5 half-lives, whichever is longer
6. Positive test at Screening for HIV, hepatitis B surface antigen (HBsAg) or hepatitis C antibody (HCV-Ab) or has a history of a positive result
7. History of alcohol or substance abuse in the past 12 months
8. Any condition that in the opinion of the investigator would jeopardize the subject's appropriate participation in this study
9. Cardiovascular conditions or medications associated with prolonged QT or those which predispose subjects to heart rhythm abnormalities.
10. Subjects with symptomatic cholelithiasis
11. Subjects with clinically significant abnormal findings during the Screening Period, and any other medical condition(s) or laboratory findings that, in the opinion of the Investigator, might jeopardize the subject's safety or ability to complete the study
12. Subjects who have been taking the following prior medications: pegvisomant (within the last 3 months), dopamine agonists (within the last 3 months) and pasireotide LAR (within the last 6 months)
13. Subjects taking octreotide LAR at a dose higher than 40 mg or lanreotide depot at a dose higher than 120 mg
14. Subjects who usually take octreotide LAR or lanreotide depot less frequently than every 4 weeks (e.g. every 6 weeks or 8 weeks)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2019-03-11 (Actual); Primary Completion 2020-07-15 (Actual); Study Completion 2020-08-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (11):
- United States (2):
  - Ohio State University, Columbus, Ohio
  - The Research Institute of Dallas, Dallas, Texas
- Brazil (2):
  - CETI - Centro de Estudos em Terapias Inovadoras, Curitiba
  - CPQuali Pesquisa Clinica, São Paulo
- General Hospital of Athens "Gennimatas", Athens, Greece
- Hungary (2):
  - Semmelweis University Faculty of Medicine, Budapest
  - University of Pécs Medical School, Pécs
- Endocrine, Diabetes and Research Centre, Wellington Hospital, Wellington, New Zealand
- The Centre of Postgraduate Medical Education, Warsaw, Poland
- Clinical Centre Serbia, Clinic for Endocrinology, Diabetes and Metabolic Diseases, Belgrade, Serbia
- National Institute of Endocrinology and Diabetology, Ľubochňa, Slovakia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Martin S, Bender RH, Krasner A, Marmon T, Monahan M, Nelson L. Development and evaluation of the Acromegaly Symptom Diary. J Patient Rep Outcomes. 2023 Feb 15;7(1):15. doi: 10.1186/s41687-023-00541-7. PMID 36792844

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Medically stable male and female subjects 18 to 75 years of age, inclusive, with a confirmed acromegaly diagnosis that was controlled on a stable approved dose of octreotide LAR or lanreotide depot. At a minimum, there had to be documentation available of a pituitary tumour and elevated IGF-1 in the past.
Pre-assignment Details: Medically stable male and female participants 18 to 75 years of age, with a confirmed acromegaly diagnosis that was controlled on a stable approved dose of octreotide LAR or lanreotide depot. There had to be documentation available of a pituitary tumour and elevated IGF-1 in the past.
Groups:
- Titration Period: Paltusotine, Then Randomized Withdrawal Period: Paltusotine: Titration Period started with the first dose of study drug (10mg all subjects) at V3, approximately 4 weeks after V1b when the last dose of standard acromegaly treatment was administered. Subjects who enrolled in the Titration Period did not receive any depot somatostatin receptor ligands (SRL) injections or other standard acromegaly treatment until study completion or early termination.
  At V6/W4, the study drug dose was titrated up in a blinded fashion, if the current dose was tolerated by the subject and the IGF-1 value at V4/W2 was >0.9×ULN (upper limit of normal for normal IGF-1 values for a specific age and sex). At V9/W7, the study drug was up-titrated in a blinded fashion if the current dose was tolerated by the subject and the IGF-1 value at V7/W5 was >ULN.
  Investigator confirmed the subject eligibility for an increase in study drug dose based on tolerability at V5/W3, V6/W4, V8/W6, and V9/W7. If tolerability was confirmed and IGF-1 reader determined that IGF-1 had not met adequate suppression criteria, a blinded blister card containing the appropriate higher dose was assigned at the V6/W4 and/or V9/W7. Dose increases in 10 mg increments were allowed only at V6/W4 (from 10 mg to 20 mg) and V9/W7 (from 10 mg to 20 mg, or from 20 mg to 30 mg) visits. No further up-titration was allowed. The daily dose did not exceed 30 mg.
  If eligible for randomization, the subject was randomized at V11/W10 in a blinded manner to continue the current dose of paltusotine.
- Titration Period: Paltusotine, Then Randomized Withdrawal Period: Placebo: Titration Period started with the first dose of study drug (10 mg for all subjects) at V3, approximately 4 weeks after V1b when the last dose of standard acromegaly treatment was administered. Subjects who enrolled in the Titration Period did not receive any depot somatostatin receptor ligands (SRL) depot injections or other standard acromegaly treatment until study completion or early termination.
  At V6/W4, the study drug dose was titrated up in a blinded fashion, if the current dose was tolerated by the subject and the IGF-1 value at V4/W2 was >0.9×ULN. Again, at V9/W7, the study drug was up-titrated in a blinded fashion if the current dose was tolerated by the subject and the IGF-1 value at V7/W5 was >ULN.
  The Investigator confirmed the subject was eligible for an increase in the study drug dose based on tolerability at V5/W3, V6/W4, V8/W6, and V9/W7. If tolerability was confirmed and the IGF-1 reader had determined that IGF-1 had not met adequate suppression criteria, a blinded blister card that contained the appropriate higher dose was assigned at the V6/W4 and/or V9/W7. Dose increases in 10 mg increments were allowed only at the V6/W4 (from 10 mg to 20 mg) and V9/W7 (from 10 mg to 20 mg, or from 20 mg to 30 mg) visits. No further up-titration was allowed. The daily dose did not exceed 30 mg.
  If determined to be eligible for randomization, the subject was randomized at V11/W10 in a blinded manner and switched to placebo.
- Titration Period: Paltusotine, Then Not Randomized: Titration period proceeded for these subjects in the same manner as other groups.
  To be eligible for randomization, the subject had to have IGF-1 value ≤ULN at V10/W8 and an Investigator determination at V11/W10 that the subject tolerated the study drug. Subjects who did not meet both criteria were not to be randomized but were to be allowed to stay in the study and continue on a study drug dose that was tolerated until completion of all study visits or until criteria to resume standard acromegaly therapy and discontinuation from the study were met. The dose of study drug used at V9/W7 remained stable through V11/W10 if tolerated.
Period: Screening Period: 4-6 Weeks
Arm/Group | Titration Period: Paltusotine, Then Randomized Withdrawal Period: Paltusotine | Titration Period: Paltusotine, Then Randomized Withdrawal Period: Placebo | Titration Period: Paltusotine, Then Not Randomized
Started | 3 | 4 | 6
Completed | 3 | 4 | 6
Not Completed | 0 | 0 | 0
Period: Titration Period: up to 9 Weeks
Arm/Group | Titration Period: Paltusotine, Then Randomized Withdrawal Period: Paltusotine | Titration Period: Paltusotine, Then Randomized Withdrawal Period: Placebo | Titration Period: Paltusotine, Then Not Randomized
Started | 3 | 4 | 6 (Titration Period lasted for up to 13 weeks for participants who did not enter the Randomized Withdrawal Period.)
Completed | 3 | 4 | 5
Not Completed | 0 | 0 | 1
Not completed — COVID-19 | 0 | 0 | 1
Period: Randomized Withdrawal: up to 4 Weeks
Arm/Group | Titration Period: Paltusotine, Then Randomized Withdrawal Period: Paltusotine | Titration Period: Paltusotine, Then Randomized Withdrawal Period: Placebo | Titration Period: Paltusotine, Then Not Randomized
Started | 3 | 4 | 5 (Non-randomized participants (who did not meet randomization criteria) did not enter the Randomized Withdrawal Period, but were allowed to stay in the study continuing on a study drug dose that was tolerated.)
Completed | 3 | 4 | 0
Not Completed | 0 | 0 | 5
Not completed — Participants who did not meet randomization criteria did not enter the Randomized Withdrawal Period. | 0 | 0 | 5
Period: Follow-up Period: up to 4 Weeks
Arm/Group | Titration Period: Paltusotine, Then Randomized Withdrawal Period: Paltusotine | Titration Period: Paltusotine, Then Randomized Withdrawal Period: Placebo | Titration Period: Paltusotine, Then Not Randomized
Started | 3 | 4 | 5
Completed | 3 | 3 | 5
Not Completed | 0 | 1 | 0
Not completed — COVID-19 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The Baseline Analysis Population includes all subjects who received treatment in the titration period. This includes subjects who were randomized in the randomized withdrawal period to receive placebo or continue receiving paltusotine and subjects who were not randomized and continued receiving paltusotine. The primary endpoint is presented for all subjects. Secondary endpoints are presented only for the randomized subjects as the RW baseline was not applicable to the non-randomized subjects.
Groups:
- Titration Period: Paltusotine, Then Randomized Withdrawal Period: Paltusotine: During the titration period, the study drug dose was titrated up in a blinded fashion. At randomization for the randomized withdrawal period, these subjects continued to receive paltusotine at the same level as end of the titration period.
- Titration Period: Paltusotine, Then Randomized Withdrawal Period: Placebo: During the titration period, the study drug dose was titrated up in a blinded fashion. At randomization for the randomized withdrawal period, these subjects were switched to placebo.
- Total: Total of all reporting groups
Arm/Group | Titration Period: Paltusotine, Then Randomized Withdrawal Period: Paltusotine | Titration Period: Paltusotine, Then Randomized Withdrawal Period: Placebo | Titration Period: Paltusotine, Then Not Randomized | Total
Number analyzed (Participants) | 3 | 4 | 6 | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 4 | 4 | 9
  >=65 years | 2 | 0 | 2 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.0 (3.00) | 38.8 (8.66) | 57.7 (11.48) | 53.5 (13.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3 | 6
  Male | 1 | 3 | 3 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 2 | 3
  Not Hispanic or Latino | 2 | 4 | 4 | 10
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 3 | 4 | 5 | 12
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Other | 0 | 0 | 1 | 1
UGT1A1 Genotype [Count of Participants; unit: Participants] — Blood sample for genotyping was analyzed for randomized subjects only and was collected for the determination of the UGT1A1 genotype. Subjects could opt out of this testing. Subjects are reported by genotype sequence (allele UGT1A1*1/*1, *1/*80, or *80/*80).
  Individuals who inherit certain polymorphisms in the UGT1A1 gene have reduced enzymatic activity. UGT1A1*1 is associated with normal enzyme activity. UGT1A1*1/*80 is associate with intermediate metabolizer phenotype and UGT1A1*80/*80 is associated with poor metabolizer phenotype
  Participants
    *1/*1 | 1 | 2 | 2 | 5
    *1/*80 | 2 | 1 | 2 | 5
    *80/*80 | 0 | 1 | 1 | 2
    Not reported | 0 | 0 | 1 | 1
UGT1A1 Phenotype [Count of Participants; unit: Participants]
  Normal Metabolizer | 1 | 2 | 2 | 5
  Intermediate Metabolizer | 2 | 1 | 2 | 5
  Poor Metabolizer | 0 | 1 | 1 | 2
  Not reported | 0 | 0 | 1 | 1
Height [Mean (Standard Deviation); unit: cm] | 163.07 (8.100) | 181.90 (14.461) | 167.73 (12.502) | 171.02 (13.748)
Weight [Mean (Standard Deviation); unit: kg] — Population: All demographics and baseline characteristics presented are based on the titration period baseline.
  kg | 70.83 (15.942) | 89.05 (10.120) | 80.65 (22.542) | 80.97 (18.088)
BMI [Geometric Mean (Standard Deviation); unit: kg/m2] — Population: All demographics and baseline characteristics presented are based on the titration period baseline.
  kg/m2 | 26.37 (3.371) | 26.95 (1.760) | 28.48 (7.008) | 27.52 (4.903)
Ring Size [Mean (Standard Deviation); unit: Scores on a Scale] — Finger size is an objective measure of soft tissue over-growth and is assessed using the US Ring Size Scale. Measurements are assessed on an increasing scale of US ring sizes scored from 1-17 (smallest to largest), with an increase in ring size between consecutive visits representing increased peripheral swelling. Ring sizers (Tool jewelry sizing tools) were provided to the sites, and sites were instructed to use the same hand and finger at each visit. Population: All demographics and baseline characteristics presented are based on the titration period baseline.
  Scores on a Scale | 13.7 (3.51) | 14.5 (5.45) | 11.3 (1.86) | 12.8 (3.63)

OUTCOME MEASURES:

1. Primary Outcome: Responder Criteria Was Based on the Mean of Two Consecutive Insulin-like Growth Factor-1 [IGF-1] Measurements ≤ULN at Week 13
Description: Proportion of subjects who meet responder criteria (based on the mean of two consecutive IGF-1 measurements ≤ upper limit of normal [ULN])
Time Frame: 13 Weeks
Population: The Analysis Population includes all subjects who received treatment in the titration period. This includes subjects who were randomized in the randomized withdrawal period to receive placebo or continue receiving paltusotine and subjects who were not randomized and continued receiving paltusotine. The primary endpoint of the proportion of subjects who met responder criteria (based on the mean of two consecutive IGF-1 measurements ≤ULN) at Week 13 is presented for all subjects.
Measure: Number (95% Confidence Interval); unit: percentage of responders
Groups:
- Randomized Withdrawal Period: Paltusotine: Subjects receiving paltusotine during the Randomized Withdrawal Period (RWP):
  Eligibility for randomization into the RWP was made based on information at the V10/W8 and V11/W10. To be eligible for randomization, the participant had to have IGF-1 value ≤ULN at V10/W8 and an Investigator determination at V11/W10 that the participant tolerated the study drug. The participants were randomized at V11/W10 in a blinded manner to continue receiving paltusotine at the same level as end of titration period.
- Randomized Withdrawal Period: Placebo: Subjects receiving placebo during the Randomized Withdrawal Period (RWP):
  Eligibility for randomization into the RWP was made based on information at the V10/W8 and V11/W10. To be eligible for randomization, the participant had to have IGF-1 value ≤ULN at V10/W8 and an Investigator determination at V11/W10 that the participant tolerated the study drug. The participants were randomized at V11/W10 in a blinded manner to be switched to a placebo.
- Randomized Withdrawal Period: Not Randomized: To be eligible for randomization, the subject had to have IGF-1 value ≤ULN at V10/W8 and an Investigator determination at V11/W10 that the subject tolerated the study drug. Subjects who did not meet both criteria were not to be randomized but were to be allowed to stay in the study and continue on a study drug dose that was tolerated until completion of all study visits or until criteria to resume standard acromegaly therapy and discontinuation from the study were met. The dose of study drug used at V9/W7 remained stable through V11/W10 if tolerated.
Arm/Group | Randomized Withdrawal Period: Paltusotine | Randomized Withdrawal Period: Placebo | Randomized Withdrawal Period: Not Randomized
Number analyzed (Participants) | 3 | 4 | 6
percentage of responders | 66.7 [9.4 to 99.2] | 25.0 [0.6 to 80.6] | 16.7 [0.4 to 64.1]

2. Secondary Outcome: Change in IGF-1 Levels
Description: Change in IGF-1 levels between RWP Baseline/Week 10 and Week 13
Time Frame: From Week 10 to Week 13
Population: Analysis Population includes all subjects who met protocol pre-specified criteria for randomization into paltusotine/placebo. Per the study design, Randomized Withdrawal Period (RWP) baseline only applies to those subjects who met criteria for randomization. RWP baseline is undefined for non-randomized subjects. Demographics and Baseline Characteristics were reported for all subjects at Titration Period Baseline, but not RWP baseline.
Measure: Mean (Standard Deviation); unit: percent change in IGF1
Arm/Group | Randomized Withdrawal Period: Paltusotine | Randomized Withdrawal Period: Placebo | Randomized Withdrawal Period: Not Randomized
Number analyzed (Participants) | 3 | 4 | 0
percent change in IGF1 | 4.04 (5.064) | 48.17 (41.408) |

3. Secondary Outcome: Change in Growth Hormone (GH) Levels
Description: Change in growth hormone levels between RWP Baseline/Week 8 and Week 13
Time Frame: From Week 8 to Week 13
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent change in GH
Arm/Group | Randomized Withdrawal Period: Paltusotine | Randomized Withdrawal Period: Placebo | Randomized Withdrawal Period: Not Randomized
Number analyzed (Participants) | 3 | 4 | 0
percent change in GH | 71.96 (48.865) | 108.30 (179.977) |

4. Secondary Outcome: Change in Total ASD Score Between RWP Baseline/Week 10 and Week 13
Description: Measured by total Acromegaly symptom diary (ASD) score from W10-W13.
  ASD is a sponsor-developed daily diary to assess important acromegaly symptoms from the patient perspective. It covers 7 symptoms (headache pain, joint pain, sweating, fatigue, weakness in legs, swelling, and numbness or tingling). Patients rate the severity of each experience in the past 24 hours on an 11-point numeric scale that ranges from 0 (no symptom) to 10 (worst symptom).
  A weekly average ASD score is calculated for each item as the sum of the item responses for a specific item over the course of the study week divided by the number of days on which the item was completed.
  The weekly average ASD total score is calculated by computing the sum of the weekly average item scores for the 7 items (total range from 0 to 70), where higher score = higher symptom severity.
Time Frame: From Week 10 to Week 13
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Total ASD score change -units on a scale
Arm/Group | Randomized Withdrawal Period: Paltusotine | Randomized Withdrawal Period: Placebo | Randomized Withdrawal Period: Not Randomized
Number analyzed (Participants) | 3 | 4 | 0
Total ASD score change -units on a scale | 1.571 (3.1004) | 7.962 (7.1591) |

ADVERSE EVENTS:
Time Frame: Duration of participation for each subject after obtaining a signed informed consent was up to 23 weeks.
Description: Safety analysis set: All participants enrolled in the study who received any amount of the study drug. All AEs reported in ≥ 1 subject are presented.
Groups:
- Safety Analysis Set/Titration Period - Paltusotine: All participants who received a dose of Paltusotine during the titration period.
- Randomized Withdrawal Period - Paltusotine: Adverse events reported during the randomised withdrawal period by those receiving Paltusotine treatment
- Randomized Withdrawal Period - Placebo: Adverse events reported during the randomised withdrawal period by those receiving Placebo
- Total Paltusotine: All participants who received a dose of paltusotine. Includes all participants randomized into the RWP, and those not randomized that were allowed to stay in the study and continue dosing at a study drug dose that was tolerated, until the participant completed all study visits.
Arm/Group | Safety Analysis Set/Titration Period - Paltusotine | Randomized Withdrawal Period - Paltusotine | Randomized Withdrawal Period - Placebo | Total Paltusotine
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/3 | 0/4 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/3 | 0/4 | 0/13
Other Adverse Events (participants affected / at risk) | 8/13 | 3/3 | 4/4 | 10/13
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Safety Analysis Set/Titration Period - Paltusotine (N=13) | Randomized Withdrawal Period - Paltusotine (N=3) | Randomized Withdrawal Period - Placebo (N=4) | Total Paltusotine (N=13)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Blood glucose increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Blood triglycerides increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 3 (3) | 1 (1) | 0 (0) | 4 (4)
Paraesthesia (Nervous system disorders) | 2 (2) | 0 (0) | 1 (1) | 2 (2)
Fatigue (General disorders) | 2 (2) | 1 (1) | 0 (0) | 3 (3)
Peripheral swelling (General disorders) | 2 (2) | 0 (0) | 1 (1) | 3 (3)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Sleep disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Due to small sample size, a number of exploratory endpoints were defined but not summarised. All primary and secondary endpoints are reported.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that PIs cannot publish until the multi-center publication is first published. If no multi-center publication is published within 18 months of the completion date, the PI may publish their results, provided that the Sponsor is given the opportunity to review the proposed publication in advance.

DOCUMENTS (2):
  • Study Protocol (2019-06-06): https://cdn.clinicaltrials.gov/large-docs/55/NCT03792555/Prot_000.pdf
  • Statistical Analysis Plan (2020-09-08): https://cdn.clinicaltrials.gov/large-docs/55/NCT03792555/SAP_001.pdf